CLINICAL TRIAL: NCT01539577
Title: A Long-Term Safety Study of OZURDEX® in Clinical Practice
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 206207-025
Record Dates: First submitted 2012-02-22; First posted 2012-02-27 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Retinal Vein Occlusion; Macular Edema; Uveitis, Posterior
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema; Uveitis, Posterior | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OZURDEX®: OZURDEX® (dexamethasone 700 μg intravitreal implant) administered according to general clinical practice.
  Interventions: Drug: dexamethasone 700 μg intravitreal implant

INTERVENTIONS:
Drug: dexamethasone 700 μg intravitreal implant — dexamethasone 700 μg intravitreal implant administered according to general clinical practice.
  Other Names: OZURDEX®

SUMMARY:
This study is a multicenter, prospective, observational study to evaluate the long-term safety of OZURDEX® in patients with macular oedema following central retinal vein occlusion (CRVO) or branch retinal vein occlusion (BRVO) or patients with non-infectious posterior segment uveitis in real-world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Macular oedema following either BRVO or CRVO or non-infectious uveitis
* Requires treatment with OZURDEX®

Exclusion Criteria:

* Current participation in any clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with macular oedema due to CRVO or BRVO or non-infectious uveitis
Sampling Method: Non-Probability Sample
Enrollment: 875 (Actual)
Dates: Start 2012-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Patients Reporting Serious Adverse Events | 2 years
Incidence of Patients Reporting Ophthalmic Adverse Events of Special Interest | 2 years
  The ophthalmic adverse events of special interest include: increased intraocular pressure, glaucoma, ocular hypertension, cataract formation and progression, vitreous detachment, haemorrhage, endophthalmitis (infectious/ non-infectious), retinitis secondary to reactivation of latent viral or other ophthalmic infections, retinal tear/detachment, significant vitreous leak or hypotony, systemic corticosteroid effects, and mechanical failure of device and implant misplacement.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (4):
- Paris, France
- Ulm, Germany
- Barcelona, Spain
- Bradford, West Yorks, United Kingdom